CLINICAL TRIAL: NCT01598129
Title: Exploratory Open Label Study of GM-CSF Coding Oncolytic Adenovirus CGTG-102, With Low Dose Cyclophosphamide in Patients With Refractory Injectable Solid Tumours
Brief Title: ONCOS-102 (Previously CGTG-102) for Therapy of Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Targovax Oy (Industry)
Responsible Party: Sponsor
Organization: Targovax ASA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oncos-C1
Record Dates: First submitted 2012-04-19; First posted 2012-05-15 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Solid Tumour
Keywords: Phase I; Dose escalation; oncolytic virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CGTG-102 (Experimental): CGTG-102 dose escalation
  Interventions: Genetic: ONCOS-102

INTERVENTIONS:
Genetic: ONCOS-102 — GMCSF encoding 3/5 chimeric adenovirus for intratumoral and intravenous injection on day 1, 4, 8, 15, 29, 57, 85, 113 and 141 tested in three different dose cohorts (3x10E10, 1x10E11 and 3x10E11) in combination with low-dose metronomic cyclophosphamide.

SUMMARY:
The purpose of the study is to investigate the safety and the recommended dose for later use of an oncolytic adenovirus CGTG-102 in combination with low-dose oral cyclophosphamide in the treatment of advanced cancers.

DETAILED DESCRIPTION:
CGTG-102 is an adenovirus that has been armed with granulocyte-macrophage colony stimulating factor (GMCSF), a potent stimulator of immunological cells.

With regard to oncolytic viruses, replication in normal cells does not take place, and therefore viruses such as CGTG-102 are not known to cause any disease. Further, to date there has been no incidence of passing the virus on to other humans from patients. Since the virus requires tumor cells to multiply, such events are unlikely.

To this day more than 100 patients have been treated with CGTG-102. This clinical trial will take place over approximately 6 months. The study includes 12 visits to the hospital, 1 screening visit, 9 injection visits including overnight stay at the hospital(performed on trial days 1, 4, 8, 15, 29, 57, 85, 113 and 141), 1 end of treatment visit (day 169) and 1 end of study visit (day 190). Oral treatment with cyclophosphamide (1 pill per day) will start on the day after the first injection and last until visit day 169.

ELIGIBILITY:
Inclusion Criteria:

1. Solid tumour refractory to evidence-based oncological therapies.
2. Age 18 years and over.
3. At least one tumour mass measurable by PET (i.e. PET-positive lesion that can reliably be assessed for SUVmax, typically featuring longest diameter ≥2 cm).
4. Tumour is injectable i.t. by direct visualisation/palpation or by imaging-guidance (ultrasound). I.t. includes intracavitary injections, particularly intraperitoneal and intrapleural.
5. Histological confirmation of primary disease or relapse.
6. Patient has given signed informed consent.
7. WHO performance score 0-1 and life expectancy more than 3 months.
8. Previous anti-cancer treatment at least 1 month before Day 1.
9. Tumour assessed to be suitable for biopsy.
10. Hepatic, renal and bone marrow functions within normal limits for the target population as indicated by the following:

    * Total bilirubin ≤ the upper limit of normal (ULN).
    * ASAT, ALAT ≤3.0 × ULN.
    * Serum creatinine ≤1.5 x ULN.
    * International normalised ratio (INR) ≤1.5 x ULN.
    * Haematologic parameters: Patients can be transfused to meet the haemoglobin and platelet count entry criteria.

      * Haemoglobin ≥10 g/dL
      * Leucocytes ≥2.3 x 109/L
      * Platelet count ≥7.5 x 109/L

Exclusion Criteria:

1. Use of high dose systemic immune suppressive medication within 3 weeks of anticipated first treatment. Note: patients taking low-dose corticosteroids for the treatment of nausea and/or taking maintenance corticosteroids are permitted to enrol.
2. Known infection with HIV or known underlying genetic immunodeficiency disease as these might affect the safety and efficacy of treatment.
3. Treatment of the injected tumour(s) with radiotherapy, chemotherapy, surgery, or an investigational drug within 4 weeks prior to the first treatment.
4. Recent thromboembolic event (deep venous thrombosis, pulmonary embolism).
5. Clinically significant active infection or clinically significant medical condition considered high risk for investigational new drug treatment (e.g. pulmonary, neurological, cardiovascular, metabolic, clinically significant and/or rapidly accumulating pericardial effusion).
6. Severe or unstable cardiac disease.
7. Known brain metastases, glioma. Central nervous system malignancy, including carcinomatosis meningitis.
8. Pulse oximetry oxygen saturation <90% at rest in room air.
9. Vaccination with a live virus (i.e. measles, mumps, rubella, etc.) <30 days prior to the first treatment.
10. History of hepatic dysfunction, cirrhosis or hepatitis.
11. Prior organ transplant.
12. Pregnant or lactating patients.
13. Evidence of coagulation disorder.
14. Other conditions which, in the opinion of the investigator, might interfere with the study findings or represent a safety hazard for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael von Euler, MD PhD, Study Director — Oncos Therapeutics Ltd.
Locations (1):
- Docrates Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Ranki T, Pesonen S, Hemminki A, Partanen K, Kairemo K, Alanko T, Lundin J, Linder N, Turkki R, Ristimaki A, Jager E, Karbach J, Wahle C, Kankainen M, Backman C, von Euler M, Haavisto E, Hakonen T, Heiskanen R, Jaderberg M, Juhila J, Priha P, Suoranta L, Vassilev L, Vuolanto A, Joensuu T. Phase I study with ONCOS-102 for the treatment of solid tumors - an evaluation of clinical response and exploratory analyses of immune markers. J Immunother Cancer. 2016 Mar 15;4:17. doi: 10.1186/s40425-016-0121-5. eCollection 2016. PMID 26981247

RESULTS

PARTICIPANT FLOW:
Groups:
- CGTG-102: CGTG-102 dose escalation
  CGTG-102: GMCSF encoding 3/5 chimeric adenovirus for intratumoral and intravenous injection on day 1, 4, 8, 15, 29, 57, 85, 113 and 141 tested in three different dose cohorts (3x10E10, 1x10E11 and 3x10E11) in combination with low-dose metronomic cyclophosphamide.
Period: Overall Study
Arm/Group | CGTG-102
Started | 12
Completed | 3
Not Completed | 9
Not completed — Disease progression | 6
Not completed — Deterioration of WHO status to WHO 4 | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 63 [38 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  Finland | 12
Number of cancer indications [Number; unit: participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any (Serious and Non-Serious) Adverse Event Measured to Assess Safety and Tolerability.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
participants | 12

2. Secondary Outcome: To Determine the Safety, Tolerability and Adverse Event Profile of CGTG-102 With Low-dose CPO. To Obtain Preliminary Evidence of Antitumour Activity.
Description: Clinical and laboratory assessment. Response rate, disease control rate, progression free and overall survival.
Time Frame: 12 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Number of Participants With Stable Disease Status as Defined by Response Evaluation Criteria In Solid Tumors (RECIST) Evaluation Three Months After Starting CGTG-102 Treatment.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | CGTG-102
Number analyzed (Participants) | 10
participants | 4

4. Other Pre Specified Outcome: Quality of Life Using EORTC QLQ-C30.
Description: To assess the feasibility and usefulness of EORTC QLQ-C30 for possible use in later studies.
Time Frame: 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: An Immune Response to Treatment Was Assessed by Measuring a Temporary Increase in Pro-inflammatory Cytokines After Treatment Was Administrered.
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
participants | 12

6. Other Pre Specified Outcome: Number of Participants With Infiltration of CD8+ T Cells Into Tumors.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
participants | 11

7. Other Pre Specified Outcome: Number of Patients With Induction of Tumor-specific CD8+ T Cells in Peripheral Blood Monomuclear Cells.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
participants | 2

8. Primary Outcome: Recommended Phase 2 Dose by Identification of Any Dose Limiting Toxicities
Description: No Dose Limiting Toxicities were observed at any dose level.
Time Frame: 6 months
Measure: Number; unit: Dose limiting toxicities
Arm/Group | CGTG-102
Number analyzed (Participants) | 12
Dose limiting toxicities | 0

ADVERSE EVENTS:
Time Frame: Patients were followed up for Adverse Events throughout the study.
Description: There was no indication of a relationship between dose of CGTG-102 and the incidence or intensity of Adverse Events.
Arm/Group | CGTG-102
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CGTG-102 (N=12)
Duodenal obstruction and small intestinal hemorrhage (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Muscle rupture (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hypoalbuminemia and peripheral oedema (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CGTG-102 (N=12)
Pyrexia (Surgical and medical procedures) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days